CLINICAL TRIAL: NCT06604260
Title: FAPi-PET Imaging of in Vivo Fibrosis in Inflammatory Bowel Disease Patients
Acronym: PIMAFI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dalia Lartey (Other)
Responsible Party: Sponsor-Investigator, Dalia Lartey, Drs, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL82160.029.22; 2022-002751-19 (EudraCT Number)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: IBD (Inflammatory Bowel Disease); Crohn Disease (CD); Ulcerative Colitis (UC)
Keywords: FAPI; fibroblast activation protein; FAP; FAPi-scan; 68Ga-FAPi PET-CT
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IBD patients (Experimental): Ulcerative colitis and Crohn's disease patients
  Interventions: Diagnostic Test: 68Ga-FAPi-46

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPi-46 — 68Ga FAPi PET-CT scan
  Other Names: FAPi-scan

SUMMARY:
Our main objective is to evaluate the feasibility of 68Ga-FAPi PET/CT in detecting intestinal fibrosis in patients with IBD. To this end, we will determine 68Ga-FAPi uptake in IBD in relation to cellular FAP expression in intestinal biopsies and resection specimens.

ELIGIBILITY:
Inclusion Criteria:

Group 1

- Adults ≥18 years with confirmed diagnosis of Crohn's disease

AND one of the following:

* Gastrointestinal complaints such as diarrhea, bloody and/ or lose stools and abdominal pain, or obstructive symptoms.
* Increased CRP (>5 mg/L) and/or fecal calprotectin levels (>250 mg/kg)
* Active disease confiremed by endoscopy ( endoscopic SES-CD score >3)
* Active disease confirmed by IUS or MRI (bowel wall thickening, signs of active disease) Group 2
* Adults ≥18 years with confirmed diagnosis of ulcerative colitis

AND one of the following:

* Active disease confirmed by endoscopy (endoscopic Mayo score ≥ 2) or
* Active disease confirmed by intestinal ultrasound (BWT > 3 mm in atleast one bowel segment and atleast one other pathological IUS parameter)
* Increased CRP (>5 mg/L) and/or fecal calprotectin levels (>250 mg/kg)

Exclusion Criteria:

* Pregnancy
* Unable to provide informed consent
* IBD-related surgeries < 5 years in medical history
* Colorectal carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of areas with increased 68Ga-FAPi uptake in Crohn's disease patients | At baseline up to week 12 of study enrolment
  Detection of areas with increased 68Ga-FAPi uptake (both visually as semi-quantitatively) in the terminal ileum and colon on baseline PET/CT of active Crohn's disease patients compared to bowel uptake reference values as derived in other Amsterdam UMC 68Ga-FAPi PET imaging studies in patients not suffering from IBD (when signed informed consent is available).
Detection of areas with increased 68Ga-FAPi uptake in ulcerative colitis patients | At baseline up to week 12 of study enrolment
  Detection of areas with increased 68Ga-FAPi uptake (both visually as semi-quantitatively) in the terminal ileum and colon on baseline PET/CT of ulcerative colitis patients compared to bowel uptake reference values as derived in other Amsterdam UMC 68Ga-FAPi PET imaging studies in patients not suffering from IBD (when signed informed consent is available).

SECONDARY OUTCOMES:
Visual and semi-quantitative evaluation of the pharmacokinetics (PK) of 68Ga-FAPi | At baseline up to week 12 of study enrolment
  Visual and semi-quantitative evaluation of the pharmacokinetics (PK) of 68Ga-FAPi in patients with a) Crohn's disease and b) ulcerative colitis compared to bowel uptake reference values as derived in other Amsterdam UMC 68Ga-FAPi imaging studies in patients not suffering from IBD (when signed informed consent is available).
Protocol optimisation | At baseline up to week 12 of study enrolment
  To define optimal (single and/or dual) time point(s) post injection for imaging FAP activity in Crohn's disease and ulcerative colitis.
Minimal tracer injection dose | At baseline up to week 12 of study enrolment
  Determine the minimal tracer injection dose required to have comparable disease detection performance on PET as to the full tracer injection dose PET.

OTHER OUTCOMES:
Correspondence 68Ga-FAPi bowel uptake conventional imaging modalities and cellular FAP | At baseline up to week 12 of study enrolment
  To determine to what extent 68Ga-FAPi bowel uptake in IBD patients corresponds to conventional imaging modalities and FAP protein and transcriptome expression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lowenberg, MD PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided